CLINICAL TRIAL: NCT00362518
Title: Vitamin C and Vitamin E Therapy in Type 2 Diabetes and Cardiovascular Risk
Brief Title: Vitamins C and Vitamin E and Cardiovascular Risk
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: David S. Schade, University of New Mexico
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 04-319; 7-04-CR-41
Record Dates: First submitted 2006-08-09; First posted 2006-08-10 (Estimated); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Diabetes
Keywords: atherosclerosis; vitamin C; vitamin E
MeSH Terms: conditions — Diabetes Mellitus; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Placebo Comparator): Study Arm A - Control: no vitamins (placebo only).
  Interventions: Dietary Supplement: Study Arm A
- 2 (Active Comparator): Study Arm B - Low Dose: Vitamin C 250 mg, Vitamin E 200 IU
  Interventions: Dietary Supplement: Study Arm B
- 3 (Active Comparator): Study Arm C - Medium Dose: Vitamin C 500 mg, Vitamin E 400 IU
  Interventions: Dietary Supplement: Study Arm C
- 4 (Active Comparator): Study Arm D - High Dose: Vitamin C 1000 mg, Vitamin E 800 IU.
  Interventions: Dietary Supplement: Study Arm D

INTERVENTIONS:
Dietary Supplement: Study Arm A — Control: no vitamins (placebo only). This study will provide baseline metabolic and surrogate marker changes that are caused by the high fat meal. Study arms B, C, and D will be statistically compared to this study.
  Arms: 1
Dietary Supplement: Study Arm B — This study arm will provide information on the response of atherogenic surrogate markers to a high fat supper when a low dosage form of vitamin C is administered (250 mg) and Vitamin E (200 IU).
  Arms: 2
Dietary Supplement: Study Arm C — This study arm will provide information on the response of atherogenic surrogate markers to a high fat supper when a medium dosage form of vitamin C administered (500 mg)and Vitamin E (400 IU).
  Arms: 3
Dietary Supplement: Study Arm D — This study arm will provide information on the response of atherogenic surrogate markers to a high fat supper when a high dosage form of vitamin C is administered (1000 mg) and Vitamin E (800 IU).
  Arms: 4

SUMMARY:
The proposed study will examine the hypothesis that vitamin C and vitamin E given to type 2 diabetic individuals will provide effective anti-inflammatory, anti-thrombotic, and anti-oxidative atherosclerotic protection when administered at the optimal dose as determined by surrogate markers of inflammation, hypercoagulability, and oxidation.

DETAILED DESCRIPTION:
This American Diabetes Association research project is to determine why there are discrepant results between individual studies of Vitamin E and C in both animals and humans compared with the results obtained in large randomized human trials using Vitamin E.

Subjects: The study will enroll subjects (both men and women) with type 2 diabetes of at least six months duration. An outpatient screening test will utilize the following: a complete history and physical examination, an EKG, a urine hcG (only for women of childbearing age), and the following blood tests: CBC, Chem-20, lipid profile, hemoglobin A1C, and C-peptide stimulation test. Subjects will be excluded if they have known vascular disease, uncontrolled hypertension (>140/90 mmHg) or marked hyperlipidemia (serum low density lipoprotein > 4.1 mmol/L or serum triglycerides > 7.8 mmol/L). Eligible patients must have normal electrocardiogram tracings and normal screening test results (described above). Other important exclusion criteria are cigarette smoking, volunteers taking Coumadin, and recent use of antioxidant supplements or aspirin. All patients will provide written informed consent before enrollment as approved by the University of New Mexico Human Research Review Committee.

Surrogate Markers: Based on our preliminary data and the published medical literature, it is extremely likely that vitamins C and E will modify all three contributors to atherosclerosis: Oxidative stress, Hypercoagulability, and Inflammation. Therefore, as shown in the table above, we have included standard surrogate markers for all three of these contributors.

Specific Aim: Determine the optimal oral dose of vitamin C and vitamin E relative to the consumption of an atherogenic high fat supper in type 2 diabetic individuals. These data are necessary in order to design prospective clinical trials in which vitamins are given to prevent or delay atherosclerotic events. One reason that published clinical trials demonstrate conflicting results may be the different dosages of vitamins that have been utilized. In the following study, we will utilize our high fat (simulated Big Mac) meal to assess the beneficial effects of these vitamins on surrogate markers of atherosclerosis. Three dosages of vitamins will be utilized in order to determine the optimal dosage.

The three dosages to be tested are 1) low dose - vitamin C 250mg, vitamin E 200 IU 2) medium dose - vitamin C 500 mg, vitamin E 400 IU and 3) high dose - vitamin C 1000mg, vitamin E 800 IU. The results will be compared to a control meal study in which only placebo (hence, no vitamins) is administered. The vitamins will be administered before breakfast on each study day.

ELIGIBILITY:
Inclusion Criteria:

* The study will enroll subjects, both men and women with type 2 diabetes of at least six months duration. The age of enrolled subjects will range from 21-60 years old. An HbA1c blood test must show that the person's diabetes is under control. Eligible subjects must have normal electrocardiogram tracings and normal hematological, electrolyte and liver laboratory results at screening. Females of childbearing age must agree to use an effective form of birth control throughout the study period.

Exclusion Criteria:

* Subjects will be excluded if they have known vascular disease, uncontrolled hypertension (>140/90 mmHg), marked hyperlipidemia (serum low density lipoprotein > 4.1 mmol/L or serum triglycerides > 7.8 mmol/L), and a body mass index greater than 40 kg/m2 (range 27-40). Other important exclusion criteria are cigarette smoking, volunteers taking Coumadin, and recent use of antioxidant supplements or aspirin. Females who are pregnant or breastfeeding will be excluded. People cannot participate in this study if they are taking medications (other than antidiabetic medications) which may affect blood sugar.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-07 (Actual); Primary Completion 2007-06 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
The goal is to determine the effects of the vitamin C and vitamin E on surrogate markers of atherosclerosis following an atherogenic meal in type 2 diabetes | 2 months

SECONDARY OUTCOMES:
To determine changes in surrogate markers of atherosclerosis in type 2 diabetes | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: David S Schade, M.D., Principal Investigator — University of New Mexico School of Medicine
Locations (1):
- University of New Mexico Health Sciences Center, Albuquerque, New Mexico, United States

REFERENCES:
- [Derived] Gutierrez AD, de Serna DG, Robinson I, Schade DS. The response of gamma vitamin E to varying dosages of alpha vitamin E plus vitamin C. Metabolism. 2009 Apr;58(4):469-78. doi: 10.1016/j.metabol.2008.11.003. PMID 19303966